CLINICAL TRIAL: NCT02736279
Title: Measuring the Impact of Tecfidera on the Gut Microbiota: Does a Change in the Gut Flora Correlate With Gastrointestinal Disturbances Following Therapy Initiation?
Brief Title: Impact of Tecfidera on Gut Microbiota
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Virginia Simnad (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor-Investigator, Virginia Simnad, MD, M.Sc, EvergreenHealth
Organization: EvergreenHealth (Other)
Other Study IDs: VIS2014
Record Dates: First submitted 2016-03-22; First posted 2016-04-13 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dimethyl fumarate — Observation of impact of dimethyl fumarate treatment initiation on mood and gut microbiome over the first 6 months of therapy
  Other Names: Tecfidera

SUMMARY:
Objectives: Dimethyl fumarate (DMF) therapy may cause a measureable change in bacterial species of the gut. The primary objectives of this study are:

1. Determine whether a measureable change in bacterial species representation follows the institution of DMF.
2. Determine whether a specific pattern of change in the microbiota phylotype with DMF therapy correlates to onset and severity of gastrointestinal disturbances (heartburn, nausea, flatulence, and diarrhea).
3. Determine whether any instability of microbiota phylotype representation persists following the institution of DMF or whether stabilization relates to resolution of gastrointestinal disturbances.
4. Determine whether there is a correlation between a pre-existing functional bowel disorder and development or severity of gastrointestinal disturbances and of peripheral eosinophilia.

Design: Double-blinded, prospective, single-center pilot study.

Patient Population: Individuals 18 years or older, with a confirmed diagnosis of a relapsing form of multiple sclerosis.

Treatment Groups: This study will be an open-label prospective study design with respect to MS immunomodulatory therapy choice. Study group will be defined as subjects with a relapsing form of multiple sclerosis, as defined by the McDonald criteria, choosing to begin DMF therapy.

DETAILED DESCRIPTION:
This will be an open-label prospective study design with respect to MS immunomodulatory therapy choice. Study group will be defined as subjects with a relapsing form of multiple sclerosis as defined by the McDonald criteria choosing to begin dimethyl fumarate (DMF) therapy. Blinding of the principal investigator and study subject to microbiota analysis results will be maintained until the planned end of study. Subjects who receive at least one dose of DMF and subsequently discontinue therapy will be invited to complete the study on alternative immunomodulatory therapy or no therapy. Data from subjects who have received at least one dose of DMF and who withdraw early from the study will be included in analysis as last visit carried forward. A goal has been set to enroll 25 subjects for this study.

Gut microbiota will be characterized using a commercial service, Second Genome, utilizing bacterial DNA extraction from stool samples and 16S ribosomal RNA gene amplification, followed by high-throughput sequencing. Taxonomic profiling on the Illumina MiSeq system is cycled to generate paired 250-bp reads in Second Genome's protocols. These longer read lengths provide high-quality full length-reads of the gene to ensure the most accurate classification available through sequencing technologies. Next generation sequencing has emerged as a powerful tool for investigating microbial communities in large sample sets.

Serial stool samples will be collected from each subject, and sent to Second Genome for analysis. The first stool sample will be collected prior to the initial dose of DMF, with subsequent collections at defined time points over the course of the study. A more intensive analysis will focus on the first 12 weeks of treatment, a time during which development and resolution of gastrointestinal side effects typically take place on therapy. Treatment-emergent flushing severity will be recorded during this time using a 5-point Likert scale flushing severity survey. Gastrointestinal (G.I.) symptoms will be assessed using the Gastrointestinal Symptoms Rating Scale (GSRS) questionnaire, a validated, self-administered questionnaire that includes 15 questions, which assess severity of G.I. symptoms using a 7-point Likert scale in five domains: indigestion, diarrhea, constipation, abdominal pain and reflux. The severity of symptoms reported in the GSRS increases with increasing score. Other variables which potentially may alter the gastrointestinal microbiota and secondarily DMF tolerance will be assessed, including the identification of subjects predisposed to functional bowel disorders via use of the Rome III functional bowel survey, a validated clinical tool to identify at-risk individuals, diet composition, antibiotic exposure, steroid treatments for neurological relapses, use of prebiotic , probiotic, or vitamin D supplements, and H2 blocker or proton pump inhibitor (PPI) therapy, as gut pH changes impact the gut flora composition.Additional data on mood change over 24 weeks of DMF therapy, using the Hamilton Anxiety Measurement (HAM) Rating Scale and Patient Health Questionnaire-9 (PHQ-9) Depression Scale, will be collected and correlated to DMF-emergent G.I. disturbances, and to changes in bacterial and archaeal species in the gut flora.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of a relapsing form of multiple sclerosis by McDonald criteria.
* Age 18 years or older.
* Able to provide informed consent.
* Treatment naïve to DMF, Fumaderm or other fumarate containing compound.
* Neurologically stable within 4 weeks prior to screening.
* Stable gross diet composition type (Western, vegetarian with dairy, vegan, gluten-limited, Paleo) within 12 weeks of screening visit.
* Able to complete study specific questionnaires and demographic information via HIPAA compliant secure internet based portal.
* No oral antibiotics within 4 weeks of screening.
* Able to abide by safety surveillance monitoring and management as part of standard of care.
* Able and willing to comply with the protocol requirements for the duration of the study.

Exclusion Criteria:

* Treatment with immunosuppressive therapies (other than steroids) within 12 months of screening, experimental or FDA approved cell trafficking modulators, experimental immune cell vaccines, or stem cell therapy.
* G.I. diagnostic or therapeutic procedure within 24 weeks of screening visit, or at any time during participation in the study.
* Steroid therapy (oral or intravenous) within 4 weeks of screening visit.
* Chronic use of a proton pump inhibitor therapy (daily use for greater than 4 weeks) within 3 months of screening.
* Chronic use (i.e. daily use for greater than 4 weeks) of laxatives other than Colace within 6 months of screening.
* Intravenous antimicrobial therapy within 24 weeks of screening.
* Oral antimicrobial therapy within 4 weeks of screening.
* Dental procedure within 4 weeks of screening visit.
* Total parenteral nutrition (TPN) within 12 months of screening.
* History of Crohns disease, ulcerative colitis, biliary cirrhosis, celiac disease, chronic pancreatitis, gastric lap-band procedure, gastric or colon cancer, bowel resection, colitis within past 6 months.
* Women who are pregnant, breastfeeding, planning pregnancy, or potentially fertile and not willing to abide by effective contraception while being treated with DMF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from a single center located in Seattle, Washington. Eligibility will be determined following a clinical decision to begin dimethyl fumarate therapy for a relapsing form of multiple sclerosis. Study population will reflect the local community composition, which is predominantly Caucasian.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Measure change in the diversity and relative abundance of bacterial and archaeal species in the gut microbiota following the start of DMF therapy. | Weeks 0 (baseline), 4,8,12,and 24
  16S ribosomal RNA gene sequencing for taxanomic classification of both known and unknown bacteria. This method quantifies the relative abundance of bacterial and archaeal species at each time point of sampling, and changes in the composition of species at specified time points from baseline (weeks 0, 4, 8, 12, and 24 following DMF treatment initiation.

SECONDARY OUTCOMES:
Measure change in anxiety level within the first 6 months following the start of dimethyl fumarate therapy. | Weeks 0 (baseline), 12, and 24
  Prospective analyses of anxiety severity comparing the aggregate score from the Hamilton Anxiety Measurement (HAM) at baseline visit prior to the start of DMF therapy to the aggregate score obtained at weeks 0 (baseline prior to therapy), 12 and 24.
Measure change in depression level within the first 6 months following the start of dimethyl fumarate therapy. | Weeks 0 (baseline), 12, and 24
  Prospective analyses of depression severity comparing the aggregate score from the Patient Health Questionnaire-9 (PHQ-9) Depression Scale survey at baseline visit (week 0) prior to the start of DMF therapy to the aggregate score obtained at weeks 12 and 24 from start of therapy.
Define pre-existing functional bowel disturbance as a predictor of GI symptoms development and severity following the start of dimethyl fumarate treatment. | Weeks 0 (baseline); 1-12 and 24
  Baseline functional GI disturbances will be quantified by the Rome III functional bowel survey prior to initiating dimethyl fumarate therapy (week 0). Following treatment initiation, developing gastrointestinal symptoms and their severity will be measured by the Gastrointestinal Symptoms Rating Scale at selected time points (weekly for the first 12 weeks, and at week 24) within the first 6 months of DMF treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia I Simnad, MD, Principal Investigator — EvergreenHealth
Locations (1):
- EvergreenHealth MS Center, Kirkland, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of all data analysis and submission of an abstract or article to a peer reviewed journal or professional meeting, each study subject may receive a copy of the aggregate data on their gut microbiome analyses from the study coordinator